CLINICAL TRIAL: NCT05941273
Title: A Study of the Implantable Miniature Telescope, Model SING (SING IMT) in Patients With Central Vision Impairment Associated With End-stage Age Related Macular Degeneration in an Israeli Cohort
Brief Title: A Study of the SING IMT in an Israeli Cohort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VisionCare, Inc. (Industry)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDV-SNG 001
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy
Keywords: Implantable Miniature Telescope
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: Single site case series
Masking Description: As the IMT has a unique appearance in the eye, it cannot be masked to the Investigator or to the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted Eye with SING IMT (Experimental): The SING IMT is implanted in on eye and safety endpoints are aimed at following that eye over time post-implant
  Interventions: Device: smaller incision, new generation implantable miniature telescope (SING-IMT)

INTERVENTIONS:
Device: smaller incision, new generation implantable miniature telescope (SING-IMT) — The IMT (model SING) is an intraocular implant comprised of 2 micro lenses in a glass tube (optics) in a flexible silicone carrier (haptics)

SUMMARY:
The objective of this single center study is to determine the safety of the smaller incision, new generation (SING), implantable miniature telescope (IMT) in a small sample of patients with moderate-severe central vision loss due to late-stage age-related macular degeneration (AMD) in an Israeli Cohort

DETAILED DESCRIPTION:
The SING IMT has CE Mark in the EU and has been implanted in over 200 patients globally including a pivotal study in the U.S. currently underway (the Concerto Study) and a post-marketing study in EU (The PMCF Study). Model SING is a new injectable model based on the IMT parent model (PMA P050034). Following completion of informed consent, patients will be evaluated for eligibility to enroll into the study, including assessment of their best-corrected distance- and near- visual acuity with refraction, and also when using an external telescope simulator to determine if they are likely to benefit from receiving the SING IMT. If eligible, they will be scheduled for out-patient surgery to implant the IMT during routine cataract surgery in one eye. Following implantation, patients will return for 5 post-operative follow-up visits over a period of approximately 12 months. Additionally, patients will have up to 10 rehabilitation/training visits with a low vision specialist to learn how to use the fellow eye for ambulation and the eye with the implant for magnified viewing during daily activities.

ELIGIBILITY:
Inclusion Criteria:

For Both Eyes:

* Be at least 55 years of age at the Pre-operative Visit;
* Have ETDRS BCDVA 0.6 to 1.6 logMAR (20/80 to 20/800) at the Pre-operative Visit;
* Have bilateral retinal findings of geographic atrophy or disciform scar with foveal involvement, as determined by fluorescein angiography (FA) or OCT;
* Have an Endothelial Cell Density (ECD) above 1800 cells per millimeter;
* Have central anterior chamber depth (ACD) >2.5 mm from the posterior surface of the cornea (endothelium) to the anterior surface of the crystalline lens at the Pre-operative Visit;
* Agree to participate in post-operative visual training

For the Implanted Eye:

* Have evidence of visually significant cataract at the Pre-operative Visit;
* Agree to undergo pre-operative assessment with low vision specialists (optometrist, occupational therapist or other professional with low vision experience) in the use of an external telescope model sufficient for patient assessment and patient must achieve at least a 5-letter ETDRS BCDVA improvement (0.1 logMAR) in the final assessment

For the Non-Implanted Eye:

-Have adequate peripheral vision at the Pre-operative Visit to allow navigation.

Exclusion Criteria:

For Both Eyes:

* Have cognitive impairment that would interfere with the ability to understand and provide Informed Consent or prevent proper visual training/rehabilitation with the device;
* Have evidence of bilateral active choroidal neovascularization (CNV) on fluorescein angiography or OCT or were treated for CNV within the past six months.
* Have any of the following conditions at the Pre-operative Visit:

  1. Stargardt macular dystrophy;
  2. Diabetic retinopathy;
  3. Untreated retinal tears;
  4. Retinal vascular disease;
  5. Optic nerve disease;
  6. History of retinal detachment;
  7. Intraocular tumor;
  8. Retinitis pigmentosa;
  9. History of steroid-induced rise in intraocular pressure (IOP), uncontrolled glaucoma, or IOP >22 mmHg at the Pre-operative Visit;
* Have known allergy to post-operative medications;
* History of eye rubbing or an ocular condition that predisposes subject to eye rubbing;
* Have had prior or expected ophthalmic surgery within 30 days of the Operative Visit;
* Have any circumstance that, based on the Investigator's judgment, poses a concern for the subject's safety;
* Any systemic disease or clinical evidence of any condition at the Pre-operative Visit which would make the subject in the opinion of the investigator unsuitable for the study;
* Concurrent participation or prior participation in any investigative drug or device study within last 30 days prior to Pre-operative Visit.

For the Implanted Eye:

* Have a history of corneal stromal or endothelial dystrophies, including guttata;
* Have Myopia > 6.0 D or Hyperopia > 4.0 D by Manifest Refraction at the Pre-operative Visit;
* Have an Axial Length (AL) < 21 mm at the Pre-operative Visit;
* Have a narrow angle defined as < grade 2 on the Schaffer scale at the Pre-operative Visit;
* Ongoing Inflammatory ocular disease at the Pre-operative Visit;
* Zonular weakness/instability of crystalline lens, or pseudoexfoliation at the Pre-operative Visit;
* Have any condition at the Pre-operative Visit which in the judgement of the Investigator indicates that the haptics cannot be placed within the capsular bag during surgery;
* Have had previous intraocular or corneal surgery, including any type of surgery for refractive or therapeutic purposes;

For the Non-Implanted Eye:

-Have ophthalmic pathology at the Pre-operative Visit that compromises the patient's peripheral vision based on the Investigator's judgment.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Endothelial cell density | Comparison of baseline to Visit 5 (330 to 420 days post-operatively)
  Percent change in endothelial cell density (ECD) from Pre-operative Visit in study

SECONDARY OUTCOMES:
Adverse Events | Approximately 12-months post-operatively (330-420 days)
  Rates of adverse events from Operative Visit through Visit 5

CONTACTS AND LOCATIONS:
Overall Officials: Guy Kleinman, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No